CLINICAL TRIAL: NCT05591950
Title: Übersetzung Und Validierung Einer Deutschen Version Der Intensive Care Unit Mobility Scale (IMS) Translation and Validation of the Intensive Care Unit Mobility Scale (IMS)
Brief Title: Translation and Validation of the Intensive Care Unit Mobility Scale (IMS)
Acronym: TAVIMS
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Stefan J Schaller, Deputy Clinical Director, Charite University, Berlin, Germany
Other Study IDs: TAVIMS
Record Dates: First submitted 2022-08-17; First posted 2022-10-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Muscle Weakness; Critical Illness; Mechanical Ventilation Complication; Early Mobilization
Keywords: ICU-mobility-scale
MeSH Terms: conditions — Muscle Weakness; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Intensive care unit acquired weakness (ICUAW) is a common issue in critically ill patients. Early mobilization can reduce the occurrence of ICUAW. This requires a standardized procedure based on validated scales. One such scale is Carol Hodgson's ICU Mobility Scale (IMS).

The subject of the study is the translation of the IMS into German and the validation of its reliability and predictive power with regard to various clinical outcomes. Furthermore we want to investigate the communication about the mobilisation status of ICU-patients between the different medical disciplines that are involved in patient care.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill adults (age: ≥ 18 years)
* Expected length of stay in ICU > 24h
* Ventilation support

Exclusion Criteria:

* Patients transferred from other ICUs
* Patients with pre-existing functional limitations
* Patients with functional limitations due to the admission diagnosis (e.g. stroke. with hemiparesis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes intensive care patients who are treated by the Clinic for Anesthesiology with focus on surgical intensive care medicine at the Charité - Universitätsmedizin Berlin for an expected period of more than 24 hours, who are at least 18 years old and receive ventilation support.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Predictive validity of the IMS | approximate 28 days (till ICU discharge)
  Predictive validity of the IMS-score performed in the first 24 hours after admission to the ICU for the length of stay in the ICU

SECONDARY OUTCOMES:
ICU mortality | approximate 28 days (till ICU discharge)
  Mortality during ICU stay
Duration of mechanical ventilation | approximate 28 days (till ICU discharge)
  Duration of invasive mechanical ventilator dependency
Discharge location | approximate at 28 days (at hospital discharge)
  If the patient was discharged home or to another facility at hospital discharge
MRC Score | approximate 28 days (till ICU discharge)
  Muscle strength at ICU discharge measured using the Medical Research Council score
Muscle strength | approximate 28 days (till ICU discharge)
  Muscle strength at ICU discharge measured using hand grip strength
90-day mortality | at 90 days
  Mortality at 90 days
90-day function | at 90 days
  Physical function of the patient at 90 days
IMS during the ICU stay | approximate 28 days (till ICU discharge)
  achieved mobilization level during the ICU stay using the ICU Mobility Scale (IMS)
ICU-LOS | approximate 28 days (till ICU discharge)
  Length of stay in the ICU
Hospital LOS | approximate 28 days (till discharge)
  Length of stay in the hospital
in-hospital mortality | approximate 28 days (till discharge)
  Mortality during the Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Univiversitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data can be requested on reasonable scientific request.
Supporting Information: Study Protocol, ICF
Time Frame: After publication of scientific manuscript.
Access Criteria: Deidentified data can be requested on reasonable scientific request.